CLINICAL TRIAL: NCT04245488
Title: Sour Taste Intensity Matching With Fatty Acids Taste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Richard Mattes, Professor, Purdue University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1901021644
Record Dates: First submitted 2020-01-23; First posted 2020-01-29 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Fat Taste

STUDY DESIGN:
Intervention Model Description: sensory
Masking Description: used three random numbers and covered cups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- taste testing (Other): Participants will first taste 5 sour solution containing acetic acid for sour compounds, sucrose esters, and xanthan gum to help them stay dissolved). Then rate them for their taste intensities. Next, participants will taste 5 butyric acid solutions, 5 hexenoic acid solutions, 5 caprylic acid solutions, 5 lauric acid solutions, 5 palmitic acid solutions, 5 oleic acid solutions, and 5 linoleic acid solutions (all will also contain the sucrose esters and xanthan gums.) and rate them for their taste intensities. This should take no longer than 1 hour. Participants will spit all samples into a cup after tasting them. They will not swallow any samples.
  Interventions: Other: taste test

INTERVENTIONS:
Other: taste test — rate intensity of sour solutions and fatty acid solutions

SUMMARY:
Investigators are trying to find the concentrations of fatty acids ( a part of the fat and flavor typically found in normal foods) that have a taste intensity similar to that to the sourness of vinegar solutions.

DETAILED DESCRIPTION:
Participants will first taste 5 sour solution containing acetic acid for sour compounds, sucrose esters, and xanthan gum to help them stay dissolved). Then rate them for their taste intensities. Next, participants will taste 5 butyric acid solutions, 5 hexenoic acid solutions, 5 caprylic acid solutions, 5 lauric acid solutions, 5 palmitic acid solutions, 5 oleic acid solutions, and 5 linoleic acid solutions (all will also contain the sucrose esters and xanthan gums.) and rate them for their taste intensities. This should take no longer than 1 hour. Participants will spit all samples into a cup after tasting them. They will not swallow any samples.

ELIGIBILITY:
Inclusion Criteria:

* male and female age 18 to 65

Exclusion Criteria:

* taste abnormalities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Intensity | 2 hours
  Participants will first taste 5 sour solution containing acetic acid for sour compounds, sucrose esters, and xanthan gum to help them stay dissolved). Then rate them for their taste intensities. Next, participants will taste 5 butyric acid solutions, 5 hexenoic acid solutions, 5 caprylic acid solutions, 5 lauric acid solutions, 5 palmitic acid solutions, 5 oleic acid solutions, and 5 linoleic acid solutions (all will also contain the sucrose esters and xanthan gums.) and rate them for their taste intensities. Rating between weak and intense.

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No